CLINICAL TRIAL: NCT03420885
Title: Ba Duan Jin for Patients With Pulmonary Nodules on Physical Condition, Psychological Condition and Quality of Life: A Pilot Clinical Study
Brief Title: Effects of Ba Duan Jin for Patients With Pulmonary Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Yueyang Integrated Medicine Hospital (Other); Longhua Hospital (Other)
Responsible Party: Principal Investigator, Lu Ying, MM, assistant researcher, Shanghai University of Traditional Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016YSN31
Record Dates: First submitted 2018-01-07; First posted 2018-02-05 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Nodules
Keywords: Ba Duan Jin; Pulmonary Nodules; Clinical Intervention
MeSH Terms: conditions — Multiple Pulmonary Nodules

STUDY DESIGN:
Intervention Model Description: A total of 60 patients were divided into a treatment group and a control group, with 30 cases in each group. The control group received health education，and the treatment group was treated with Ba Duan Jin plus health education program.
Who Masked: Outcomes Assessor
Masking Description: The study was a single-blind controlled trial in which the outcome assessor was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ba Duan Jin Group (Experimental): Ba Duan Jin plus health education. Participants take part in 16-week program. The health education is conducted as the Health Education Group. Besides, the participants attended two 90-minute sessions of group-based Ba Duan Jin training per week and practiced at least three 30-minute Ba Duan Jin sessions at home per day.
  Interventions: Behavioral: Ba Duan Jin; Behavioral: Health Education
- Health Education Group (Active Comparator): Health education. Participants take part in 16-week program. The health education includes work, rest, diet and other basic programs according to the different conditions of participants.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Ba Duan Jin — Ba Duan Jin, a traditional Chinese health-preserving technique, combines the traditional Chinese medicine and traditional Chinese philosophy and embrace the body, breath and spirit. Ba Duan Jin consists of eight main movements. According to traditional theory, every movement has unique effect to different Zang-fu organs.
  Other Names: Eight-section Brocade
  Arms: Ba Duan Jin Group
Behavioral: Health Education — Health education includes work, rest, diet and other basic programs according to the different conditions of participants.

SUMMARY:
Many researches shows that Ba Duan Jin has clinical efficacy on cancer rehabilitation, respiratory diseases, psychological health, quality of life and so on. Studies examining the effects of Ba Duan Jin on patients with pulmonary nodules are sparse. Therefore, the aims of the present study are: 1) to examine the effects of Ba Duan Jin on physical and psychological condition, and 2) to examine the effects of Ba Duan Jin on quality of life.

DETAILED DESCRIPTION:
In recent years, with advancement in computed tomography (CT) technology and its widespread use, pulmonary nodules are common incidental findings. Pulmonary nodules are used to appear as well-circumscribed radiographic opacity. They can be single or multiple. There are multiple causes of pulmonary nodules. Most nodules are benign, but some may also represent bronchogenic carcinoma or metastatic lesions. The prevalence of malignancy is detected nodules varies between 0.2% and 18%. Thus, the preoperative individuals would suffer from depression or anxiety caused by uncertain progression of pulmonary nodules; the postoperative individuals would suffer from both physical and mental trauma.

There is growing interest in non-pharmacological approaches that could potentially improve pulmonary nodules patients' physical condition, psychological condition and quality of life.

Ba Duan Jin, a traditional Chinese health-preserving technique, combines the traditional Chinese medicine and traditional Chinese philosophy and embrace the body, breath and spirit. There is substantial evidence that Ba Duan Jin has benefits for cancer rehabilitation, respiratory diseases, psychological health, and quality of life. The effects of Ba Duan Jin on patients with pulmonary nodules are yet to be further investigated.

The present pilot clinical study aims to apply Ba Duan Jin to patients with pulmonary nodules, and to evaluate the effects on physical (pulmonary function), psychological (depression and anxiety), and quality of life. Participants allocated to the Health Education Group take part in the 16-week health education including work, rest, diet and other basic programs according to the different conditions of participants. Participants allocated to the Ba Duan Jin Group take part in the 16-week Ba Duan Jin plus health education program. The study plans to enroll 60 participants in 2 years (30 for Ba Duan Jin plus health education program, and 30 for health education program), expecting that Ba Duan Jin has a better effect on improving physical condition, psychological condition and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed by CT scan of the lung(s).
* Subject is male or female, age 18 to 75.
* Subject has a clear mind and the ability to read, to talk and to communicate.
* Subject agrees to participate in this study and sign to the informed consent.

Exclusion Criteria:

* Subject has recurrence of cancer.
* Subject has severe somatic disease.
* Subject has history of psychosis, mania, or severe personality.
* Subject is pregnant, lactating or breast-feeding women.
* Subject is engaging in other clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-18 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Vital Capacity in liters (VC) | 16 weeks
  VC, a measure of pulmonary function, is the maximum amount of air a person can expel from the lungs after a maximum inhalation.
Forced Vital Capacity in liters (FVC) | 16 weeks
  FVC, a measure of pulmonary function, is the volume of air that can forcibly be blown out after full inspiration.
Forced Expiratory Volume in one second in liters (FEV1) | 16 weeks
  FEV1, a measure of pulmonary function, is the volume of air that can forcibly be blown out in one second, after full inspiration.
FEV1/FVC in percents (FEV1%) | 16 weeks
  FEV1% is the ratio of FEV1 to FVC.
Peak Expiratory Flow in liters (PEF) | 16 weeks
  PEF, a measure of pulmonary function, is the maximal flow (or speed) achieved during the maximally forced expiration initiated at full inspiration.
the Zung Self-Rating Anxiety Scale (SAS) | 16 weeks
  The SAS, designed by Duke University psychiatrist William W.K. Zung MD, is a 20-item self-report assessment built to measure anxiety level. Each items points accumulated as raw score, then the raw score will be converted into a percentage (the SAS index); the higher the SAS index, the greater the severity of anxious symptoms.
the Zung Self-Rating Depression Scale (SDS) | 16 weeks
  The SDS, designed by Duke University psychiatrist William W.K. Zung MD, is a 20-item self-report assessment built to measure depression level. Each items points accumulated as raw score, then the raw score will be converted into a percentage (the SDS index); the higher the SDS index, the greater the severity of depressive symptoms.

SECONDARY OUTCOMES:
the MOS 36-Item Short Form Health Survey(SF-36) | 16 weeks
  The SF-36 is a 36-item, patient-report survey of patient health status. It consists of eight scaled scores and each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. Higher scores indicate a better health-related quality of life.
CT scan of the Lung(s) | 16 weeks
  Follow-up CT scan imaging is required to observe the changes of pulmonary nodules in size, density, type and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lu, Study Director — Shanghai Qigong Research Institute
Locations (1):
- Shanghai Qigong Research Institute, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu Y, Li J, Ni W, Li J, Song J, Jiang J, Zhao X. Effectiveness of mind-body exercise via Baduanjin on physical and psychological outcomes in patients with pulmonary ground-glass nodules: A non-randomized controlled pilot study. Complement Ther Clin Pract. 2023 Feb;50:101679. doi: 10.1016/j.ctcp.2022.101679. Epub 2022 Nov 9. PMID 36399997